CLINICAL TRIAL: NCT02449499
Title: Interpersonally Focused Psychodynamic Group Psychotherapy as Adjunct Treatment for Residual Symptoms of Major Depressive Disorder
Brief Title: Adjunct Interpersonally Focused Psychodynamic Group Psychotherapy for Residual Depression Symptoms
Status: Terminated | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Carrie Holmberg, protocol director, Stanford University
Other Study IDs: IRB-32272
Record Dates: First submitted 2015-04-07; First posted 2015-05-20 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- therapy: patients who meet inclusion criteria, continue to work with individual therapist, and participate in adjunct weekly group therapy
- control: patients who meet inclusion criteria, continue to work with individual therapist, and are eligible for group therapy participation but cannot participate in group due to schedule constraints

SUMMARY:
Depression and anxiety disorders, even when treated according to standard of care consisting of individual treatment with medication and/or therapy, can be associated with significant residual impact on quality of life. The purpose of this research is carry out an observational study of an existing clinical treatment, adjunctive interpersonally focused psychodynamic group therapy, to determine if this can improve quality of life for patients who have residual symptoms of chronic depression and anxiety.

DETAILED DESCRIPTION:
Patients will be referred from primary individual therapist at the Stanford psychiatry outpatient clinics or community. Patients meeting inclusion criteria will be contacted for consent to participate in intake process consisting of objective evaluation with Patient Health Questionnaire (PHQ9; assessment of mood), Generalized Anxiety Disorder Scale (GAD7; assessment of anxiety), Psychological General Well-Being Index (PGWBI), adult attachment style questionnaire (ASQ), and the interpersonal communication inventory (ICI), followed by standardized interpersonally oriented intake interview. Test and interview administration will be done by resident psychiatrists with training by supervising psychiatry faculty. A Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) diagnosis will be obtained using the Mini-International Neuropsychiatric Interview (MINI). Patients entered on antidepressants will be held at a stable dosage. Patients will be required to continue to see their individual therapist throughout the duration of their participation in the study, and will be asked for consent for group leaders to speak with individual therapist as clinically indicated.

A total of 25 patients are projected to be entered into the group. Rolling enrollment will proceed to maintain a minimum of 5 and maximum of 10 people in the group, as expected group therapy drop-out rates are on the order of 30%. This number of people is expected to provide sufficient group membership for effective interpersonal psychodynamic group therapy. The group will use psychodynamic principles tailored to the group setting, which focus on interpersonal dynamics happening within the group in real-time, as described in Dr. Irvin Yalom's Group Psychotherapy text. Sessions will be 75 minutes in length on a weekly basis. Sessions will be led by two senior (4th year) psychiatry residents and videotaped for supervision by two faculty psychiatrists. During the study, all group members will complete PHQ9, GAD7, and Sheehan disability scale prior to each group therapy session. The full battery of objective assessments delivered at the start of the study will be repeated every 6 months. Study will involve group participation for six months, with the option to continue in the group afterwards. Subjects who withdraw prior to 6 months will be asked to complete the full battery of objective assessments otherwise administered every 6 months and their data will be used as pilot data examining outcomes at intermediary time points.

Additionally, age and gender matched patients who meet inclusion criteria but are unable to attend group sessions due to scheduling conflict will be given objective scales described above at screening and at 6 months (or earlier if clinical or treatment status changes). This group will act as control. They will continue to engage in their typical individual psychiatric care, as the goal of this study is to examine additional benefit of adjunct group therapy above individual therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* MINI diagnosis of major depression, adjustment disorder, generalized anxiety disorder, panic disorder, social phobia, or depression not otherwise specified (NOS)
* PHQ9 <20 and/or GAD7>5 despite minimum of 6 months of prior psychiatric treatment
* Poor interpersonal, social, academic, work or home function based on clinical assessment and subjective self-report
* Effective engagement with group therapy task as assessed during standardized initial screening which is to demonstrate a willingness and ability to engage in an effective therapeutic manner with others in the group
* Ongoing treatment by primary individual psychotherapist
* Insurance with behavioral health coverage accepted at Stanford clinics

Exclusion Criteria:

* Active serious medical conditions
* Traumatic Brain Injury (TBI), dementia, developmental delay or severe cognitive impairment
* Psychotic or substance abuse issues
* On newly prescribed psychiatric medication <30 days on stable target dose
* Currently in acute depressive episode
* Personality disorder
* Suicidality
* Inability to speak/understand English fluently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with major depression, adjustment disorder, generalized anxiety disorder, panic disorder, social phobia, or other depression NOS diagnosis currently in treatment with individual psychotherapist, continuing to experience symptoms even after at least six months in standard individual treatment with a psychiatrist or psychologist.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-04; Primary Completion 2015-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
psychological and general well-being index | 6 months

SECONDARY OUTCOMES:
ASQ (adult attachment style questionnaire) | 6 months
ICI (interpersonal communication inventory) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Holmberg, MD, PhD, Principal Investigator — Stanford Psychiatry and Behavioral Science
Locations (1):
- Stanford Psychiatry and Behavioral Science, Palo Alto, California, United States